CLINICAL TRIAL: NCT02072811
Title: Evaluation of the Efficacy of Induction-consolidation Treatment Using a Double Induction in Patients With AML <60 Years Old, Depending on the Percentage of Blasts in the 14 Day, Residual Disease and Leukemic Hematopoietic Cells
Brief Title: Role of the Therapy Tailored to Risk Factors in Treating Adult Patients (≤60) With Acute Myeloid Leukemia
Acronym: PALG-AML2012
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: dr hab. n. med. Agnieszka Wierzbowska (Other)
Collaborators: Polish Adult Leukemia Group (Other); Copernicus Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, dr hab. n. med. Agnieszka Wierzbowska, PhD in Copernicus Memorial Hospital, Hematology Department, Polish Adult Leukemia Group
Organization: Polish Adult Leukemia Group (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALG-AML2012
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Daunorubicin; Granulocyte Colony-Stimulating Factor; Mitoxantrone; 2'-chloro-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Induction, DAC (Other): The first stage of treatment.
  First DAC induction cycle is common to all patients (regardless of risk group). After completion of induction I occurs early assessment of bone marrow on the +14 day after the start of treatment (+7 day after completion of chemotherapy).
  Interventions: Drug: DAC
- II early induction, CLAG (Other): Patients with blasts in the bone marrow in D14> 10% receive early second induction (CLAG) which start form +16 day.
  Patients with blasts in the bone marrow in D14 ≤ 10% do not receive early second induction and are qualified to assess the response times on +28 day or after full morphology recovery (if it occurs before the +28 day
  Interventions: Drug: CLAG
- Consolidation, I HAM cycle (Other): I induction cycle starts after complete remission (CR).
  - After I consolidation, patients from Intermediate I an Intermediate II group (ELN prognostic system):
  If compatible donor is present - allogeneic HSCT qualification after I or II consolidation. If compatible donor for allogeneic HSCT is not present - attempt to CD34+ mobilization for autologous SCT after II consolidation
  - After I consolidation, patients from Adverse risk group (ELN prognostic system):
  If compatible donor is present - immediate qualification for allogeneic HSCT.
  - Finding a donor should be initiated in all patients, at the latest after the end of I induction. In the first place, it should be checked whether the patient has a donor family, if not - searching start for an unrelated donor. For patients with no compatible donor for allogeneic HSCT - need to start searching for an alternative donor
  Interventions: Drug: Consolidation, I HAM cycle
- II Consolidation HiDAraC (Other): Patients from all 5 risk group receive second after first consolidation [Ara-C] Patient from Very adverse risk receive Ara-C + CLA (Cladribine). If it is needed - more intensive consolidation treatment with 2-Cda.
  Patients form Very adverse risk receive Maintenance treatment:
  Decitabine 20 mg/m2 60 min infusion iv (Intravenous injection) for 5 days every 6 weeks.
  Patients from Favorable, - Intermediate I an Intermediate II risk groups: CD34+ mobilization (HSCT qualification).
  Interventions: Drug: II Consolidation HiDAraC
- Consolidation, III HiDAraC cycle (Other): Patients from Favorable, Intermediate I an Intermediate II risk groups receive III consolidation or autologous HSCT (depends on results of mobilization).
  Patients from Adverse risk receive III Consolidation HiDAraC + Cladribina (CLA) If no CR: CLAG-M reinduction therapy and after CR - treatment according to protocol.
  Interventions: Drug: Consolidation, III HiDAraC cycle

INTERVENTIONS:
Drug: DAC — * DNR 60 mg/m2 0,5h infusion iv on 1-3 days
  * 2-CdA 5 mg/m2 2h. infusion iv on 1-5 days
  * Ara-C 200 mg/m2 12h infusion iv 2h after end of infusion with 2CdA on 1-7 days
  Other Names: - Cladribine; - Cytosine arabinoside [Ara-C]; - Daunorubicin
  Arms: Induction, DAC
Drug: CLAG — * G-CSF 30MU sc, on 0-5 days
  * Mitoxantrone 10mg/m2 30 min infusion iv, on 1-3 days
  * Cladribine 5mg/m2 in 2h infusion iv, on 1-5 days
  * Ara-C 2000mg/m2 4h infusion iv, infusion start after 2h of Cladribine infusion end, on 1-5 day
  Other Names: - Granulocyte-colony stimulating factor [G-CSF]; - Cladribine; - Mitoxantrone; - Cytosine arabinoside [Ara C]
  Arms: II early induction, CLAG
Drug: Consolidation, I HAM cycle — * Ara-C 3g/m2; 3h infusion iv every 12h on 1,2,3 days
  * Mitoxantrone 10mg/m2; 0,5h infusion iv on 3,4,5 days
  Other Names: - Mitoxantrone; - Cytosine arabinoside [Ara-C]
  Arms: Consolidation, I HAM cycle
Drug: II Consolidation HiDAraC — • Ara-C 3g/m2 every 12h; 3h infusion iv on 1,3,5 days (+ mobilization of CD34+)
  Other Names: - Cytosine arabinoside [Ara-C]; - Cladribine
  Arms: II Consolidation HiDAraC
Drug: Consolidation, III HiDAraC cycle — * Ara-C 3g/m2 every 12h; 3h infusion iv on 1,3,5 days
  * 2-CdA 5 mg/m2 2h infusion iv on 1,3,5 days, 2h before Ara-C
  Other Names: - Cytosine arabinoside [Ara-C]; - 2-CdA [Cladribine, 2-Chlorodeoxyadenosine]
  Arms: Consolidation, III HiDAraC cycle

SUMMARY:
In view of the diversity of the biology of acute myeloid leukemia (AML) therapy in individual patients must be individualized. One of the tools for this is molecular-cytogenetic stratification. It divides patients into five categories (prognostic groups): Favorable, Intermediate-1, Intermediate-2, Adverse and Very adverse risk. After remission proceedings are tailored depending on prognostic determined groups.

Research of PALG group in the application in the second line regimen CLAG and CLAG-M proved high effectiveness of this treatment with low toxicity. Considering experience of PALG groups, it seems that the use of the schema CLAG early as the second induction therapy is a viable treatment option.

DETAILED DESCRIPTION:
Patients with AML with one of 5 prognostic categories based on modified cytogenetic-molecular stratification (European Leukemia Net Prognostic System - ENL)

Favorable risk

t(8;21)(q22;q22); RUNX1-RUNX1T1 inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11 Mutated NPM1 without FLT3-ITD (NK) Mutated CEBPA (NK)

Intermediate I risk

Mutated NPM1 with FLT3-ITD (NK) Wild-type NPM1 and FLT3-ITD (NK) Wild-type NPM1 without FLT3-ITD (NK)

Intermediate II risk

t(9;11)(p22;q22); MLLT3-MLL cytogenic abnormalities other than favorable or adverse

Adverse risk

Inv(3)(q21q26.2) or t(3;3)(q21;q26.2); RPN-EVI1

Very adverse risk monosomal karyotype (MK): -5 or del(5q); -7; abnl(17p); complex karyotype

Goals:

* Evaluation of the impact of therapy tailored to the risk factors on outcome of AML patients aged ≤ 60.
* Evaluation of the possibility to improve the results of induction therapy through the use of early 2nd induction in patients with persistent leukemic infiltration of the bone marrow at the 14th day,
* Evaluation of the impact of the minimal residual disease (MRD) presence assessed by Immunophenotyping method, on the results of treatment of AML patients aged ≤ 60,
* Assessing the significance of monitoring the number of leukemic stem cells (LSC) in bone marrow and peripheral blood and their influence on clinical course and outcome of AML treatment,
* Assessment of the LSC determination usefulness in MRD monitoring in patients with AML,
* Evaluation of the prognostic significance of the expression of CXCR-4 on the surface of leukemic cells and their impact on the clinical course and outcome of AML - trying to select a group of patients who potentially would benefit from the use of chemosensitization with plerixafor,
* Evaluation of autologous HSCT effectiveness in consolidation therapy in AML patients from 3 following cytogenetic-molecular risk groups: Favorable, Intermediate I, Intermediate II,
* Comparison of the overall survive (OS) and leukemia-free survival after autologous and allogeneic HSCT in AML patients from Intermediate I and Intermediate II cytogenetic-molecular risk groups (biological randomization donor vs. donor).

ELIGIBILITY:
Inclusion Criteria:

* Adult acute myeloid leukemia
* Age: ≥18 and ≤ 60
* Clinical condition of the patient allows to carry out induction therapy: ECOG performance status: ≤ 2 and the Hematopoietic Cell Transplant-Co-morbidity Index (HCT-I): ≤3
* Informed consent to participate in the study (ICF signed)
* The second early induction start criteria is in addition to the listed above, the percentage of the blasts on the level >10% on 7th day.

Exclusion Criteria:

* No informed consent for participation in the study, mental illness, which don't allow to obtain informed consent and conduct the treatment according to the protocol
* Pregnancy
* HIV infection
* Active cancer
* Active hepatitis virus infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Complete remission after induction | 28 days
  Outcome measure after induction:
  At +28 day after treatment or after full morphology recovery (if it occurs before the +28 day)
  Complete remission, according to Cheson's CR criteria:
  * Lack of extramedullary infiltration,
  * Platelet count> 100 G / L,
  * Neutrophil count> 1.0 G / L,
  * Lack of blast cells in the blood,
  * Bone marrow blasts <5% in the cytomorphology.
  After induction treatment, patients are qualified for one of the pro-remission treatment options, which is associated with cytogenetic-molecular risk groups, according to the modification of the molecular ELN / MDACC.
  Therapeutic decisions are being made according to cytogenetic-molecular stratification: Favorable, Intermediate-1, Intermediate-2, Adverse and Very adverse risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Copernicus Memorial Hospital, Lodz, Poland

REFERENCES:
- [Derived] Pluta A, Robak T, Brzozowski K, Stepka K, Wawrzyniak E, Krawczynska A, Czemerska M, Szmigielska-Kaplon A, Grzybowska-Izydorczyk O, Nowicki M, Stelmach P, Kuydowicz M, Gromek T, Hus M, Helbig G, Grosicki S, Bodzenta E, Razny M, Wojcik K, Bolkun L, Kloczko J, Knopinska-Posluszny W, Piekarska A, Hellman A, Sobas M, Wrobel T, Patkowska E, Lech-Maranda E, Warzocha K, Holowiecki J, Giebel S, Wierzbowska A. Early induction intensification with cladribine, cytarabine, and mitoxantrone (CLAM) in AML patients treated with the DAC induction regimen: a prospective, non-randomized, phase II study of the Polish Adult Leukemia Group (PALG). Leuk Lymphoma. 2020 Mar;61(3):588-603. doi: 10.1080/10428194.2019.1678151. Epub 2019 Oct 29. PMID 31661339